CLINICAL TRIAL: NCT02699788
Title: Emergency Department MCG for Suspected Acute Coronary Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled, sponsor refused to pay site invoices.
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TGH0006
Record Dates: First submitted 2016-02-01; First posted 2016-03-04 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multifunction Cardiogram (Experimental): non-invasive computerized, multiphase, resting electrocardiogram analysis device
  Interventions: Device: Multifunction Cardiogram

INTERVENTIONS:
Device: Multifunction Cardiogram

SUMMARY:
The goal of this study is to assess a new non-invasive computerized, multiphase, resting electrocardiogram analysis device in early identification of patients at risk for acute coronary syndrome. The overall objective is to assess the association between the results from a resting MCG and 30-day cardiovascular outcome in patients presenting to the emergency department with suspected coronary disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* Symptoms consistent with a possible acute coronary syndrome per the treating emergency physician.
* Has an electrocardiogram performed while in the ED.

Exclusion Criteria:

* Acute ST-segment elevation MI.
* Patient unable or unwilling to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Accuracy of MCG as assessed by the development of major adverse cardiac events (MACE). | 30 days
  MACE will be defined as the composite of cardiac death, myocardial infarction (MI), or coronary revascularization.
  2.2 Seco11dary

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wilson, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No